CLINICAL TRIAL: NCT06313385
Title: The Effect of Indocyanine Green Titration on Fluorescent Intensity Degree in Free Flap : A Lookout to Flap Surface Temperature, TCPO2, TCPCO2, HIF-1 Alpha Expression Level, and Histopathology
Brief Title: Investigating the Impact of Indocyanine Green Titration on Fluorescent Intensity in Free Flap : An Exploration of Alternative Indicators
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Parintosa Atmodiwirjo, Head of Center for Advanced Reconstructive Microsurgery, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 22-10-1180
Record Dates: First submitted 2024-01-15; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Free Flap; Indocyanine Green; Microsurgery; Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes | interventions — Temperature; Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Intervention Model Description: The population were divided into three equal groups of indocyanine green concentration : 5 milligram per milliliter (mg/mL), 2,5 mg/mL, and 0,5 mg/mL
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants didn't know about indocyanine green (ICG) drug groups as well as the concentration that they received. The ICG was added into the syringe by research assistant without any label near the end of operation time. The ICG injection to the patient was performed by anesthesiologist who didn't know about the concentration at all. Outcome assessor didn't know about the given concentration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 5 mg/mL (Experimental): This group received 5 mg/mL concentration of Indocyanine Green (Aurogreen®, Aurolab, Tamil Nadu, India). Indocyanine Green (ICG) is being diluted with 5 mL dextrose 5%. The research assistant take 1 mL ICG using 1 mL syringe using filter that originated from the Aurogreen package.
  Interventions: Diagnostic Test: Indocyanine Green Fluorescence (ICG); Diagnostic Test: Temperature; Diagnostic Test: Transcutaneous oxygen and carbon dioxide pressure; Diagnostic Test: Histopathology; Diagnostic Test: Hypoxia inducible factor-1 (HIF-1) alpha
- Group 2,5 mg/mL (Active Comparator): This group received 2,5 mg/mL concentration of Indocyanine Green (Aurogreen®, Aurolab, Tamil Nadu, India). Indocyanine Green (ICG) is being diluted with 5 mL dextrose 5%. The research assistant take 0,5 mL ICG using 1 mL syringe using filter that originated from the Aurogreen package. The ICG in the syringe is added with 0,5 mL Dextrose 5%.
  Interventions: Diagnostic Test: Indocyanine Green Fluorescence (ICG); Diagnostic Test: Temperature; Diagnostic Test: Transcutaneous oxygen and carbon dioxide pressure; Diagnostic Test: Histopathology; Diagnostic Test: Hypoxia inducible factor-1 (HIF-1) alpha
- Group 0,5 mg/mL (Active Comparator): This group received 2,5 mg/mL concentration of Indocyanine Green (Aurogreen®, Aurolab, Tamil Nadu, India). Indocyanine Green (ICG) is being diluted with 5 mL dextrose 5%. The research assistant take 0,1 mL ICG is taken using 1 mL syringe using filter that originated from the Aurogreen package. The ICG in the syringe is added with 0,9 mL Dextrose 5%.
  Interventions: Diagnostic Test: Indocyanine Green Fluorescence (ICG); Diagnostic Test: Temperature; Diagnostic Test: Transcutaneous oxygen and carbon dioxide pressure; Diagnostic Test: Histopathology; Diagnostic Test: Hypoxia inducible factor-1 (HIF-1) alpha

INTERVENTIONS:
Diagnostic Test: Indocyanine Green Fluorescence (ICG) — The ICG will be injected intravenously and being assessed with Near-infrared (NIR) camera FLUORO4000XL 20 cm above the flap and fluorescence intensity counted with application called ImageJ
  Other Names: ICG fluorescence
Diagnostic Test: Temperature — Portable thermal imaging camera called Forward-looking infrared (FLIR) ONE® was used to assess flap and normal skin temperature. The FLIR ONE® device was place in perpendicular manner from the skin. The images were attained in two points of times which is direct temperature and after cold challenge test.
Diagnostic Test: Transcutaneous oxygen and carbon dioxide pressure — The partial transcutaneous pressure is measured in flap using transcutaneous monitor (TCM) Combi probe. The probe should be cleaned using alcohol pads before use. After 5-10 minutes, the TCM 4 machine monitor should show stable transcutaneous oxygen and carbon dioxide pressure from the flap
Diagnostic Test: Histopathology — A part of tissue from free flap is acquired and stored in 10% formalin tube. Later on, the tissue was colored with hematoxylin-eosin, neutrophile count, necrosis volume, and vessel proliferation will be assessed
Diagnostic Test: Hypoxia inducible factor-1 (HIF-1) alpha — Peripheral tissue from distal free flap (0,5 x 0,5 cm in size) is obtained and stored in tube with dry ice. The tissue is assessed with human HIF - 1 Alpha Enzyme-Linked Immunosorbent Assay (ELISA) kit ab171577.

SUMMARY:
This study is a randomized clinical trials that aim to determine the effect of Indocyanine Green (ICG) titration dose on the intensity degree of ICG fluorescence imaging results. In addition, this study will also determine the relationship of other indicators such as flap surface temperature, transcutaneous pressure of carbon dioxide (TcPCO2), transcutaneous pressure of oxygen (TcPCO2), HIF - 1 alpha expression, and flap histopathology morphology to the intensity degree of ICG fluorescence imaging results with titrated doses.

DETAILED DESCRIPTION:
The ICG contrast solution will be evaluated with Near-Infrared (NIR) camera that being fixated 20 cm above the flap after the injection. The imaging result will be analyzed using ImageJ Application to assess the grey value. The fluorescent intensity of ICG will be compared with other tests.

Drop Out Criteria :

* Patients who are unable to complete the research procedure due to various condition, such as death
* Patients who experience complications or worsening, during and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Free flap operation that being performed by researchers.
* Free Flap must have a skin paddle located on the body skin area with intraoperative ischemic time of at least 60 Minutes
* Free flap should be in a viable/vital condition judged from the clinical examination of the flap, which includes color, temperature, turgor, capillary refill time (CRT), and skin prick test, immediately post surgery
* Body area that will be a flap-free donor area has no history of trauma or operation
* Patient with blood albumin value >3 gr / dL
* The patient/family sign the informed consent sheet stating willingness to become research sample

Exclusion Criteria:

* Patients have increased sensitivity to iodine or ICG
* Free Flaps that being transported undergo trauma or damage due to external factors during treatment
* Patient with high urea and creatinine level
* Patient with high Alanine transaminase (ALT) and Aspartate transaminase (AST) level
* Patients who receive injectable heparin treatment containing natrium disulfite preoperatively
* Patients who regularly take anti-seizure drugs, haloperidol, heroin, meperidine, Metamizole, methadone, morphine, nitrofurantoin, opium, phenobarbital, and phenylbutazone.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-03-29 (Estimated)

PRIMARY OUTCOMES:
The Effect of Indocyanine Green Fluorescence Intensity to evaluate free flap perfusion | Immediate Postoperative, 24 hours after surgery, 72 hours after surgery, 120 hours after surgery
  The fluorescence of ICG that being captured with near-infrared (NIR) camera is store in video file to be evaluated. The video duration is 2 minutes long after ICG injection. The fluorescence intensity of the flap in the video is being measured with ImageJ application. The highest level of intensity (numerical data) is considered as the optimal fluorescence intensity that being analyzed later on. The optimal indocyanine green titration will be seen after ImageJ analysis in numerical data called gray values.

SECONDARY OUTCOMES:
The ICG fluorescence intensity in different titration dose with flap surface Temperature | Immediate Postoperative, 24 hours after surgery, 72 hours after surgery, 120 hours after surgery
  The surface temperature of the flap and the surrounding normal tissue is being measured with mobile thermal camera. The temperature result is shown in celsius degree
Correlation between ICG fluorescence intensity in different titration dose with transcutaneous carbon dioxide and oxygen pressure | Immediate Postoperative, 24 hours after surgery, 72 hours after surgery, 120 hours after surgery
  The transcutaneous carbon dioxide and oxygen pressure are shown in mmHg after being measured with transcutaneous (TCM) Combi 4 device.
Correlation between ICG fluorescence intensity concentration in different titration dose with flap neutrophile count | Immediate Postoperative, 24 hours after surgery, 72 hours after surgery, 120 hours after surgery
  The neutrophile count is shown as cells per high power field. The high power field in this study is 20x optical view magnification in microscope. This is part of histopathology examination.
Correlation between ICG fluorescence intensity concentration in different titration dose with flap necrosis volume | Immediate Postoperative, 24 hours after surgery, 72 hours after surgery, 120 hours after surgery
  The necrosis volume result is shown in numerical data percentage (%). High power field which is 20x optical view magnification in microscope. This is part of histopathology examination.
Correlation between ICG fluorescence intensity concentration in different titration dose with vascular flap proliferation of the tissue | Immediate Postoperative, 24 hours after surgery, 72 hours after surgery, 120 hours after surgery
  The vascular flap proliferation can be seen using after the tissue sample is stained immunohistochemically using cluster of differentiation (CD) 31 marker in 20x optical view magnification using microscope. The result will be seen in numerical data. This is part of histopathology examination.
Correlation between ICG fluorescence intensity in different titration dose with HIF-1 Alpha | Intraoperative (before start of anastomosis and before end of anastomosis time), 24 hours after surgery, 72 hours after surgery, 120 hours after surgery
  The ICG fluorescence intensity in 3 different titration dose will be compared with HIF-1 Alpha. The HIF-1 Alpha will be shown as numerical value in ng/mg of proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Parintosa Atmodiwirjo, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Cipto Mangunkusumo Hospital, Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No